CLINICAL TRIAL: NCT02246114
Title: Self-Monitoring of Carbon Monoxide to Enhance Reproductive Outcomes in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor of Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000370
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy; Smoking; Smoking Cessation
Keywords: Pregnancy; Smoking; Smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no CO monitor (Experimental): Not given a piCO+ Smokerlyzer® monitor, will receive daily text messages.
  Interventions: Other: Text messages
- CO monitor (Experimental): Given a piCO+ Smokerlyzer® monitor, will receive daily text messages, will receive feedback about the relative level of carbon monoxide.
  Interventions: Device: piCO+ Smokerlyzer® monitor; Other: Text messages

INTERVENTIONS:
Device: piCO+ Smokerlyzer® monitor
  Arms: CO monitor
Other: Text messages

SUMMARY:
Our goal is to study self-monitoring of smoking as a means to reduce smoking in pregnant women. Investigators hypothesize that more regular self-monitoring, text messages and feedback as provided by home carbon monoxide monitoring device combined with medical feedback on results will reduce smoking during pregnancy compared to only receiving text message and no self-monitoring by home monitoring device and no feedback by home carbon monoxide monitoring device . The periconceptual period is a life period, where given the immediacy of the fetus and future child, a pregnant woman is willing to try and modify potentially harmful behaviors.

DETAILED DESCRIPTION:
Altering unhealthy behaviors, such as tobacco smoking, that increase cardiovascular disease and cancer risk, has proven remarkably difficult in traditional medical practice settings, and successful medical trials have been costly and labor intensive. This proposal aims to utilize a self-monitoring device, i.e., carbon monoxide monitor to foster smoking cessation among pregnant women who smoke. Investigators hypothesize that women who have access to a self-monitoring device more frequently (i.e., at home) and receive feedback about their carbon monoxide level will have greater reductions in smoking as determined by declining serum cotinine levels over the course of the study compared to women who do not have access to a self-monitoring device and do not receive feedback about their carbon monoxide level, but only receive text messages.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-40 years old
* Participants will be pregnant women estimated to be between 6 and 20 weeks into their pregnancy
* Pregnant women have smoked at least at least one cigarette in the prior 7 days
* Own a smartphone capable of delivering and receiving text messages

Exclusion Criteria:

* Project materials and text messages are in English, potential participants will be excluded if they cannot read English and if there are concerns about the ability to comprehend or comply with study procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- MS Hershey Medical Center, Penn State College of Medicine, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: no CO monitor
- Arm B: CO monitor
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — miscarriage | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 32 [32 to 32] |  | 32 [32 to 32]
Gender [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome of Serum Cotinine Levels
Description: The primary outcome is the difference in serum cotinine levels between the intervention and control groups at the end of the trial.
Time Frame: 1 year
Population: Only 1 subject enrolled in this study and she terminated early due to miscarriage at 9 weeks.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm A (no CO Monitor): no CO monitor
- Arm B (CO Monitor): CO monitor
Arm/Group | Arm A (no CO Monitor) | Arm B (CO Monitor)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (no CO Monitor) (N=1) | Arm B (CO Monitor) (N=0)
headache (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study closed early due to lack of recruitment. Only 1 subject enrolled in the study and she terminated after the baseline visit due to a miscarriage at 9 weeks. Therefore no analysis has been performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes